CLINICAL TRIAL: NCT00196105
Title: Multicenter Prospective Randomized Controlled Trial of the Nitinol ZILVER Expandable Endoprosthesis in the Palliation of Extrahepatic Malignant Biliary Obstruction
Brief Title: Malignant Obstruction ZILVER Against Routine Therapy (MOZART I)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-MOZ
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2010-01-12 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Biliary Tract Neoplasms; Pancreatic Neoplasms; Jaundice, Obstructive
Keywords: Stents; Stent-graft; Minimally invasive; Biliary Tract Cancer; Pancreatic Cancer; Jaundice; Biliary Tract Neoplasms; Pancreatic Neoplasms; Jaundice, Obstructive; Zilver
MeSH Terms: conditions — Biliary Tract Neoplasms; Pancreatic Neoplasms; Jaundice, Obstructive; Jaundice

ARMS (3):
- 6 mm Zilver (Experimental): 6 mm Nitinol Zilver Stent
  Interventions: Device: 6 mm Nitinol Zilver Stent
- 10 mm Zilver (Experimental): 10 mm Nitinol Zilver Stent
  Interventions: Device: 10 mm Nitinol Zilver Stent
- 10 mm Wallstent (Active Comparator): 10 mm Stainless Steel Wallstent
  Interventions: Device: 10 mm Stainless Steel Wallstent

INTERVENTIONS:
Device: 6 mm Nitinol Zilver Stent
  Arms: 6 mm Zilver
Device: 10 mm Nitinol Zilver Stent
  Arms: 10 mm Zilver
Device: 10 mm Stainless Steel Wallstent
  Arms: 10 mm Wallstent

SUMMARY:
This study compares the 6 mm nitinol Zilver biliary endoprostheses and the 10 mm nitinol Zilver biliary endoprostheses to the 10 mm Wallstent in appropriate patients in need of palliative treatment of malignant obstructive jaundice.

DETAILED DESCRIPTION:
This research is being done to determine if the new, FDA-cleared Zilver metal biliary stent is better than the conventional stents. The new Zilver stent may permit more accurate placement, may avoid some potential complications and last longer than the conventional stents. The study will also examine to find the best diameter of stent by comparing standard 10 mm stents to 6 mm Zilver stents.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable malignancy of the extrahepatic bile duct

Exclusion Criteria:

* Age below 21 years
* Pregnancy
* Active alcohol or drug abuse
* Simultaneously participating in another investigational drug or device study.
* Allergy to stainless steel or nitinol
* Active cholangitis
* Brachytherapy
* Unable or unwilling to comply with follow up

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2003-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Howell, M.D., Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

REFERENCES:
- [Result] Loew BJ, Howell DA, Sanders MK, Desilets DJ, Kortan PP, May GR, Shah RJ, Chen YK, Parsons WG, Hawes RH, Cotton PB, Slivka AA, Ahmad J, Lehman GA, Sherman S, Neuhaus H, Schumacher BM. Comparative performance of uncoated, self-expanding metal biliary stents of different designs in 2 diameters: final results of an international multicenter, randomized, controlled trial. Gastrointest Endosc. 2009 Sep;70(3):445-53. doi: 10.1016/j.gie.2008.11.018. Epub 2009 May 30. PMID 19482279

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 6 mm Zilver | 10 mm Zilver | 10 mm Wallstent
Started | 64 | 88 | 89
Completed | 60 | 83 | 82
Not Completed | 4 | 5 | 7
Not completed — Lost to Follow-up | 4 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 mm Zilver | 10 mm Zilver | 10 mm Wallstent | Total
Number analyzed (Participants) | 64 | 88 | 89 | 241
Age Continuous [Mean (Full Range); unit: Years] | 71.3 [41 to 90] | 72.8 [48 to 94] | 71.5 [49 to 96] | 71.9 [41 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 43 | 45 | 115.0
  Male | 37 | 45 | 44 | 126.0
Biliary Sphincterotomy [Number; unit: Participants]
  Patients with Biliary Sphincterotomy | 39 | 50 | 49 | 138
  Patients without Biliary Sphincterotomy | 25 | 38 | 40 | 103
Previous Plastic Stent [Number; unit: Participants]
  Patients with Previous Plastic Stent | 32 | 35 | 47 | 114
  Patients without Previous Plastic Stent | 32 | 53 | 42 | 127
Tumor Diagnosis [Number; unit: Participants]
  Patients with Pancreatic Cancer | 48 | 63 | 70 | 181
  Patients with Metastatic Cancer | 4 | 12 | 8 | 24
  Patients with Cholangiocarcinoma | 7 | 5 | 5 | 17
  Patients with Gallbladder Cancer | 1 | 0 | 2 | 3
  Patients with Other Cancer | 3 | 7 | 3 | 13
  Patients without Tumor | 1 | 1 | 1 | 3
Bilirubin [Mean (Standard Deviation); unit: mg/dL] | 9.6 (8.7) | 8.7 (7.3) | 8.3 (8.7) | 8.8 (8.2)
Karnofsky Index [Mean (Standard Deviation); unit: Units on a Scale] — The Karnofsky index runs from 100 to 0, where 100 is "perfect" health and 0 is death.
  Units on a Scale | 80.5 (9.5) | 80.6 (9.9) | 81.2 (9.2) | 80.8 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: Patency
Description: Number of days of stent patency: The time to stent occlusion requiring re-intervention, death, loss to follow-up, or patients alive at study end without an occlusion (>= 6 months after placement).
Time Frame: up to 32 months
Measure: Median (Full Range); unit: Days
Arm/Group | 6 mm Zilver | 10 mm Zilver | 10 mm Wallstent
Number analyzed (Participants) | 64 | 88 | 89
Days | 110 [7 to 595] | 125.5 [5 to 671] | 121 [0 to 961]
Statistical Analysis 1: Comparison: 6 mm Zilver vs 10 mm Zilver vs 10 mm Wallstent; Test type: Superiority or Other; p = .057, Log Rank

2. Primary Outcome: Closure or Blockage of the Stent (Occlusion)
Description: Biliary stents may become closed or blocked. This is also termed "Occlusion." Data for this outcome measure involve stent occlusions that required re-intervention.
Time Frame: up to 32 months
Measure: Number; unit: Stent Occlusions
Arm/Group | 6 mm Zilver | 10 mm Zilver | 10 mm Wallstent
Number analyzed (Participants) | 64 | 88 | 89
Stent Occlusions | 25 | 21 | 19
Statistical Analysis 1: Comparison: 6 mm Zilver vs 10 mm Zilver vs 10 mm Wallstent; Test type: Superiority or Other; p = .04, Chi-squared
Statistical Analysis 2: Comparison: 6 mm Zilver vs 10 mm Zilver vs 10 mm Wallstent; Test type: Superiority or Other; p = .007, Log Rank — Death is censored for Kaplan-Meier analysis
Statistical Analysis 3: Comparison: 10 mm Zilver vs 10 mm Wallstent; Test type: Superiority or Other; p = .69, Chi-squared
Statistical Analysis 4: Comparison: 6 mm Zilver vs 10 mm Zilver vs 10 mm Wallstent; 6 mm Zilver vs. 10 mm Zilver and 10 mm Wallstent combined; Test type: Superiority or Other; p = .02, Chi-squared — P-value is adjusted for multiple comparisons

3. Primary Outcome: Number of Days to Occlusion
Time Frame: up to 32 months
Measure: Median (Full Range); unit: Days
Arm/Group | 6 mm Zilver | 10 mm Zilver | 10 mm Wallstent
Number analyzed (Participants) | 25 | 21 | 19
Days | 115 [7 to 595] | 111 [6 to 506] | 103 [7 to 386]
Statistical Analysis 1: Comparison: 6 mm Zilver vs 10 mm Zilver vs 10 mm Wallstent; Test type: Superiority or Other; p = .16, ANOVA

4. Primary Outcome: Number of Deaths
Time Frame: up to 32 months
Measure: Number; unit: Participants
Arm/Group | 6 mm Zilver | 10 mm Zilver | 10 mm Wallstent
Number analyzed (Participants) | 64 | 88 | 89
Participants | 4 | 6 | 2

5. Primary Outcome: Time to Death
Description: Overall Survival
Time Frame: up to 32 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 6 mm Zilver | 10 mm Zilver | 10 mm Wallstent
Number analyzed (Participants) | 64 | 88 | 89
Days | 132.6 [74 to 328] | 186 [92 to 304] | 170 [99 to 273]
Statistical Analysis 1: Comparison: 6 mm Zilver vs 10 mm Zilver vs 10 mm Wallstent; Test type: Superiority or Other; p = .32, Log Rank
Statistical Analysis 2: Comparison: 6 mm Zilver vs 10 mm Zilver vs 10 mm Wallstent; Test type: Superiority or Other; p = .69, Kruskal-Wallis

ADVERSE EVENTS:
Description: No adverse events were captured due to terminal patients.
Arm/Group | 6 mm Zilver | 10 mm Zilver | 10 mm Wallstent
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days